CLINICAL TRIAL: NCT02527057
Title: Diffusion-weighted Magnetic Resonance Imaging(DW-MRI) for Early Response Assessment of Neoadjuvant Chemoradiation Therapy(Neo-CRT) in Patients With Esophageal Squamous Cell Carcinoma(ESCC)
Brief Title: Diffusion-weighted Magnetic Resonance Imaging (DW-MRI )for Early Response Assessment in Patients With Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Wang, chief of thoracic radiation oncology department, Hunan Province Tumor Hospital
Other Study IDs: 89000--0000
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Esophageal Carcinoma
Keywords: Diffusion-weighted magnetic resonance imaging; Preoperative concurrent chemoradiation; Response
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DW-MRI — Participants will perform four DW-MRI scanning as follows,before chemoradiation , at 2 weeks , 4 weeks after the start of radiotherapy and before the surgery.If participants can not receive surgery,the last scanning time will replaced at the end of radiotherapy.

SUMMARY:
Esophageal carcinoma is a lethal disease, causing more than 400,000 deaths annually worldwide. Primary surgery results in microscopically positive resection margins (R1) in 25% patients, and the 5-year overall survival(OS) for such patients rarely exceeds 40%. Concurrent chemoradiation followed by surgery results in better survival than single-modality treatments, and thus National Comprehensive Cancer Network(NCCN) recommends concurrent chemoradiation as preoperative or definitive treatment for patients with stage II or III esophageal cancer. However, neoadjuvant chemoradiation may not be effective in some subgroup of these patients, and its toxicity can increase perioperative mortality and delay or preclude surgery. The ability to distinguish tumors that will respond or not respond to such therapy remains an urgent priority. Diffusion-weighted magnetic resonance imaging(DW-MRI) is based on the extent of mobility of water protons, as quantified by the apparent diffusion coefficient (ADC). The ADC is a measure of the extent of free diffusion of water molecules within tissues, which is mainly influenced by cell organization, size, and density. Cell death leads to a loss of cell membrane integrity and density and leads to increases in ADC values. The ADC has emerged as a potential biomarker of response to cancer therapy. However, no one has published findings regarding the potential correlation between changes in ADC and response of esophageal cancer to chemoradiation. Clarifying the potential predictive value of DW-MRI for predicting response to such therapy is important for the delivery of appropriately tailored treatment.

Investigators hypothesized that DW-MRI can predict the success (or failure) of neoadjuvant chemoradiation in esophageal squamous cell carcinoma（ESCC）, hence identify patients at high risk of treatment failure from such therapy. Investigators will test this hypothesis with two specific aims: (1) assess the ability of ADC to predict pathologic response to treatment; and (2) assess the ability of ADC to predict disease-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* T1bN+ M0(T1b means that tumor invades submucosa) or T2-T4aN0/+ M0 (T4a means resectable tumor invading pleura, pericardium, or diaphragm) according to American Joint Committee on Cancer （AJCC）Cancer Stage 7th
* Pathological identified esophageal squamous cell cancer
* Karnofsky Performance Status（KPS）≥70
* Tolerable and agree for Intensity-Modulated Radiation Therapy（IMRT） and concurrent chemoradiotherapy
* Without severe other diseases
* Informed consent

Exclusion Criteria:

* Cervical esophagus cancer;
* Had received prior chemotherapy and thoracic radiotherapy
* Distant metastasis before treatment, including: pleural, pericardial or peritoneal cytology ,involvement of distant organs including the lungs, liver, bone, brain or non-regional lymph nodes
* Pregnant and lactating women
* Serious complications
* Other primary malignancies
* Cannot perform DW-MRI at specified time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will have histologically confirmed esophageal squamous cell carcinoma with no contraindications for receiving neoadjvuant chemoradiation followed by surgery. All participants will be required to give informed consent to participate in the protocol, which has been approved by the review boards of the participating institutions.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic response | after surgury
  Pathologic response will be assessed after surgery by two pathologists blinded to clinical and radiologic findings in the surgical specimen as follows : P0: no residual cancer cells P1: 1%-50% residual cancer cells; rare individual cancer cells or minute clusters of cancer cells P2: More than 50% residual cancer cells, often grossly identifiable at primary site

SECONDARY OUTCOMES:
Overall survival | up to 60 months
  Overall survival is defined as the time (in months) from the date of admission to the date of death from any cause or last follow-up
Progression free survival | up to 60 months
  Overall survival is defined as the time (in months) from the date of admission to the date of progression

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan province tumor pospital, Changsha, Hunan, China